CLINICAL TRIAL: NCT03927599
Title: Prospective and Retrospective Register Study of PARP-Inhibitors Combined With VEGFR-Inhibitors for Treatment of Advanced Refractory Solid Tumors Patients With TP53 Mutations
Brief Title: Advanced Refractory Solid Tumors With TP53 Mutations Register Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PV-TP53
Record Dates: First submitted 2019-04-22; First posted 2019-04-25 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-04

CONDITIONS: Solid Tumor, Adult
Keywords: TP53; PARP; VEGFR; Solid tumor
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Advanced refractory tumor solid tumors patients: Patients with advanced refractory solid tumors carrying TP53 mutations and receive PARP-inhibitors in combination with the VEGFR-inhibitors therapy
  Interventions: Other: Data Collection

INTERVENTIONS:
Other: Data Collection — Colleciton of data from medical records only

SUMMARY:
The efficacy and safety of the PARP inhibitor in combination with the VEGFR inhibitor will be investigated in advanced refractory solid tumors patients with TP53 mutation .

DETAILED DESCRIPTION:
TP53 is a well-known tumor suppressor gene. Multiple studies have demonstrated that TP53 mutations are poor prognostic factor in advanced solid tumor, the TP53 gene is frequently inactivated by mutation in a majority of human tumors. However, no effective TP53 -based therapy has been successfully translated into clinical cancer treatment. So, investigators intend to review and evaluate the efficacy and safety of the PARP inhibitor in combination with the VEGFR inhibitor for TP53 mutation in advanced refractory solid tumors patients from a real-world population.

ELIGIBILITY:
Inclusion Criteria:

1. Is equal to or greater than 18 years of age.
2. Histologic or cytologic confirmation of advanced refractory solid tumors with no standard treatment options, including some patients with advanced disease in reduced general condition (Eastern Cooperative Oncology Group (ECOG) 3 and 4).
3. Patients with measurable or evaluable disease per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1.
4. Patients must be able to provide blood samples or tissue samples for NGS (Next Generation Sequencing) testing for understanding the TP53 gene status. The amount of blood and tissue samples should be able to meet the requirements of DNA extraction and quality control.
5. Adequate baseline organ system function.
6. Patients could receive treatment program from MTB (Molecular Tumor Board).
7. No prior treatment with PARP combined with VEGFR inhibitions.
8. Ability to understand and the willingness to provide a written informed consent document.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding.
2. Prior anti-cancer therapy or radiation therapy within 2 weeks prior to enrolment. Palliative radiotherapy to metastatic lesion(s) permitted providing that it has been completed at least 2 days prior to enrolment and no significant toxicity are expected.
3. Clinically significant (active) cardiovascular disease: cerebral vascular accident/stroke or myocardial infarction within 6 months prior to study enrollment; unstable angina, congestive heart failure or a serious cardiac arrhythmia requiring medication.
4. Active infection requiring systemic therapy.
5. Patients unable to swallow orally administered medication.
6. Prior treatment with PARP or VEGFR inhibitions.
7. According to the investigator'judgment, there are serious, uncontrollable risks to patients'safety, or associated diseases (such as severe diabetes, thyroid disease, infection, spinal cord compression, superior vena cava syndrome, neurological or psychiatric disorders and so on) that affect the patients completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The objective is to describe in a real-world population.First of all, this study will be carried out as a retrospective, observational review of patients who clinically diagnosed as advanced refractory solid tumors received PARP-inhibitors combined with VEGFR-inhibitors drug therapy, from January 01, 2016 to August 01, 2018. The TP53 gene status must confirm by NGS (Next Generation Sequencing). Then, the investigators prospective observation effectiveness and safety of PARP-inhibitors combined with VEGFR-inhibitors therapy for patients who clinically diagnosed as advanced refractory solid tumors according to the inclusion and exclusion criteria. Those patients should have a NGS report to show the TP53 gene status.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
ORR(Objective Response Rate) | Up to three months
  ORR is the percentage of participants with best overall response of complete response (CR), partial response (PR). Response categories: CR, PR, SD (stable disease), PD (progressive disease) Criteria on which physicians determined therapy response also will be captured by using Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1 to evaluate.

SECONDARY OUTCOMES:
PFS (Progression Free Survival), calculated from various time points | Up to two years
  Progression-free survival (PFS) is defined as progression free survival of all the evaluable participants who receive targeted drug therapy. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1).
OS (Overall Survival), calculated from various time points | Duration of time from the start of treatment to date of death, assessed up to two years
  OS is defined as time from initiation to death of any cause.
ADR (Adverse Drug Reaction) | 30 days after last dose
  Adverse events determined according to CTCAE (version 4.03).

CONTACTS AND LOCATIONS:
Overall Officials: Haitao Wang, Principal Investigator — Tianjin Medical Unversity Second Hospital
Locations (1):
- Tianjin Medical Unversity Second Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided